CLINICAL TRIAL: NCT06738030
Title: Transcranial Stimulation Combined With Auditory Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7799E; R21DC021763 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Difficulties Understanding Speech in Noise
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to active transcranial stimulation or sham stimulation groups.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active transcranial stimulation (Experimental): This group will receive active transcranial alternating current stimulation that matches the envelope of the target speech.
  Interventions: Device: Transcranial current stimulation; Behavioral: Auditory training
- Sham stimulation (Sham Comparator): This group will receive transcranial stimulation that ramps on and off before the speech is presented.
  Interventions: Behavioral: Auditory training

INTERVENTIONS:
Device: Transcranial current stimulation — The transcranial alternating current stimulation is delivered during the speech stimulus and the current matches the envelope of the target speech
  Arms: Active transcranial stimulation
Behavioral: Auditory training — An at-home auditory training program that adaptively and interactively trains the listener in degraded speech, cognitive skills, and communication strategies

SUMMARY:
The goal of this clinical trial is to learn if non-invasive brain stimulation (called transcranial stimulation) can enhance the benefits from auditory training in people who struggle to understand one talker when many people are talking at the same time. The main questions it aims to answer are:

* Does transcranial stimulation improve speech-on-speech understanding in people who struggle with this task?
* Does transcranial stimulation enhance the benefits of a commercially available auditory training program?

Researchers will compare transcranial stimulation to sham stimulation (no stimulation is applied during the listening task).

Participants will:

* Receive login information to an online auditory training program to complete at home over 2 weeks
* Visit the laboratory 4 times to receive transcranial stimulation while listening to speech-on-speech: once before at-home training, two times during the at-home training period, and once after at-home training has ended

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Audiometric thresholds that do not exceed 90 dB HL at any frequency from 250-6000 Hz
* Able to provide informed consent and understand experimental instructions
* Able to read print on a computer screen
* Difficulty with speech-on-speech understanding
* Access to computer or mobile phone with access to internet that can play sound (for the at-home training)

Exclusion Criteria:

* Non-native speakers of English
* History of skull fracture, scalp tissue damage, metallic implants around the head, seizures, neurological disorders, or traumatic brain injury, current or suspected pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Speech-on-speech intelligibility percent correct | From enrollment to the end of participation at 6 weeks
  Percent correct score on the speech-on-speech task assessed in the lab
Pupillometry measured listening effort | From enrollment to the end of participation at 6 weeks
  The peak pupil dilation subtracted from pre-trial baseline pupil dilation, averaged across trials in a block, assessed in the lab
QuickSIN SNR Loss | Days 1, 6, and 14 of the two-week auditory training
  A speech-in-noise test assessed as part of the at-home auditory training program
Hearing Handicap Inventory | Days 1 and 14 of the two-week auditory training program
  A listening effort questionnaire given as part of the at-home auditory training program

CONTACTS AND LOCATIONS:
Locations (1):
- Communication Neuroscience Research Lab at Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The complete archive of all de-identified (anonymized) experimental data will be made available via Boston University's institutional archive repository "OpenBU". This will include individual participant scores on tasks and pupil dilation data. The data will be labeled with a unique study ID.
Supporting Information: Analytic Code
Time Frame: This data will be available no later than the end of the grant performance period (9/2026) and will be available indefinitely.
Access Criteria: This data will be accessible to anyone via the stable URL link managed by the BU library.